CLINICAL TRIAL: NCT07340567
Title: Tailoring the Decision for Adjuvant Chemotherapy Using Circulating Tumour DNA, in Patients With Stage III Colorectal Cancer
Brief Title: Personalizing Chemotherapy Selection After Surgery for Patients With Stage III Colorectal Cancer Using a Blood Test
Acronym: CIRCULATEIII
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Natera, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-GIG-2410
Record Dates: First submitted 2025-12-18; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine; Oxaliplatin; folfirinox; Folfox protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ctDNA-negative cohort : Capecitabine alone (Experimental): ctDNA-negative patients will be included and randomized to de-escalation treatment (capecitabine [CAPE] for 6 months).
  Interventions: Drug: Capecitabine
- ctDNA-negative cohort : Capecitabine + oxaliplatin (Active Comparator): ctDNA-negative patients will be included and randomized to standard treatment (CAPOX for 3 months).
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin
- ctDNA-positive cohort : FOLFIRINOX (Experimental): ctDNA-positive patients will be randomized to escalation treatment (5FU + irinotecan + oxaliplatin [FOLFIRINOX] for 6 months).
  Interventions: Drug: Folfirinox
- ctDNA-positive cohort : FOLFOX (Active Comparator): ctDNA-positive patients will be randomized to standard treatment (FOLFOX for 6 months).
  Interventions: Drug: FOLFOX regimen

INTERVENTIONS:
Drug: Capecitabine — De-escalation treatment (capecitabine [CAPE] for 6 months). Or Standard treatment (CAPOX for 3 months)
  Arms: ctDNA-negative cohort : Capecitabine + oxaliplatin; ctDNA-negative cohort : Capecitabine alone
Drug: Oxaliplatin — Standard treatment (CAPOX for 3 months)
  Arms: ctDNA-negative cohort : Capecitabine + oxaliplatin
Drug: Folfirinox — Escalation treatment (5FU + irinotecan + oxaliplatin [FOLFIRINOX] for 6 months)
  Arms: ctDNA-positive cohort : FOLFIRINOX
Drug: FOLFOX regimen — Standard treatment (FOLFOX for 6 months)
  Arms: ctDNA-positive cohort : FOLFOX

SUMMARY:
CIRCULATE-III is an international, multicenter, open-label, randomized phase III trial designed to use ctDNA as a selection criterion for intensification or de-escalation of adjuvant chemotherapy. Eligible patients are randomly assigned to the following treatment groups:

* Patients who test negative for ctDNA receive either capecitabine for 6 months (experimental group) or oxaliplatin + capecitabine for 3 months (standard group).
* Patients who test positive for ctDNA receive either FOLFIRINOX for 6 months (experimental group) or FOLFOX for 6 months (standard group).

Patient participation in the trial will not exceed 66 months after randomization, including a maximum treatment duration of 6 months and a follow-up period of 60 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have signed a written informed consent prior to any trial specific procedures. When the patient is physically unable to give their written consent, an impartial witness of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent
2. Age ≥18 years and <80 years (for patients aged >70 years: G8 geriatric questionnaire score>14)
3. Histologically confirmed stage III pMMR/MSS colon and high rectum adenocarcinoma (T, N1 or N2, M0) excluding medium and low rectal cancers (≥12 cm from the anal verge by endoscopy and/or above the peritoneal reflection at surgery are still eligible), without gross or microscopic evidence of residual disease after surgery with curative intent.
4. No metastatic disease on CT-Scan and/or liver MRI done within 2 months before inclusion
5. Inclusion planned between 10 days to 6 weeks after surgery
6. ECOG performance status 0-1 (fit to receive FOLFIRINOX therapy)
7. No prior chemotherapy for CRC
8. No prior abdominal or pelvic irradiation for CRC
9. Adequate hematological function: neutrophils ≥1,500 /mm3, platelet count ≥100,000/mm3, hemoglobin ≥9 g/dL (5,6 mmol/L)
10. Total bilirubin ≤1.5 x ULN (upper limit of normal)
11. ASAT and ALAT ≤2.5 x ULN
12. Alkaline phosphatase ≤2.5 x ULN
13. Serum creatinine ≤120 μmol/L or creatinine clearance ≥50 mL/min according to Modification of Diet in Renal Disease (MDRD) formulae
14. Tumor tissue available at baseline
15. Women of childbearing potential must have negative serum pregnancy test done within 7 days before the start of study treatment
16. Men and women of childbearing potential must agree to use adequate contraception methods for the duration of study treatment and for 6 months after treatment discontinuation
17. Patients must be willing and able to comply with the protocol for the duration of the study including scheduled visits, treatment plan, laboratory tests and other study procedures
18. Patient must be affiliated to a social security system (or equivalent) or according to local regulatory requirements

Exclusion Criteria:

1. Peripheral neuropathy grade ≥1
2. Patients who have received neo-adjuvant treatment.
3. Comorbidity influencing the 3-year patients' survival including clinically relevant cardiovascular disease, such as Ischemic myocardial infarction in the last year and/or unstable ischemic cardiopathy
4. Contra-indication to chemotherapy (inadequate bone marrow, hepatic, renal functions, hypersensitivity to one of the treatments or any of the excipients)
5. Patient must not have received bone marrow transplant
6. Patient must not have received blood transfusion within 3 months before inclusion
7. Participation in another therapeutic trial
8. Partial or complete dihydropyrimidine deshydrogenase (DPD) deficiency.
9. MSI/dMMR tumors
10. Medical history of other concomitant or previous malignant disease, except adequately treated in situ carcinoma of the uterine cervix, basal or squamous cell carcinoma of the skin, or cancer in complete remission for ≥ 5 years.
11. Pregnant or breastfeeding women.
12. Patients unwilling or unable to comply with the medical follow-up required by the trial because of geographic, familial social or psychological reasons
13. Persons deprived of their liberty or under protective custody or guardianship.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2450 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2032-11-01 (Estimated); Study Completion 2035-11-01 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of 6-month CAPE vs 3-month CAPOX ACT in terms of 3-year Disease Free Survival ctDNA-negative cohort | DFS will be defined as time from date of randomization until the date of first documented recurrence local or metastatic, date of second colorectal cancer, or date of death from any cause wichever came first, assessed up to 42 months.
  ctDNA-negative cohort: The primary objective is to evaluate the non-inferiority of 6-month capecitabine alone (CAPE; de-escalation strategy) compared to 3-month capecitabine + oxaliplatin (CAPOX; standard therapy) in terms of 3-year disease-free survival (DFS) as adjuvant chemotherapy (ACT) protocol in stage III pMMR/MSS CRC patients with post-operative ctDNA-negative.
Superiority of 6-month FOLFIRINOX vs 6-month FOLFOX ACT in terms of 3-year Disease Free Survival ctDNA-positive cohort | DFS will be defined as time from date of randomization until the date of first documented recurrence local or metastatic, date of second colorectal cancer, or date of death from any cause, wichever came first, assessed up to 42 months.
  ctDNA-positive cohort: The primary objective is to evaluate the superiority of 6-month FOLFIRINOX (escalation strategy) compared to 6-month FOLFOX (standard therapy) in terms of 3-year DFS as an ACT protocol in stage III pMMR/MSS CRC patients with post-operative ctDNA-positive.

CONTACTS AND LOCATIONS:
Locations (5):
- Institut Gustave Roussy, Villejuif, France
- Sweden (4):
  - Sahlgrenska University Hospital, Gothenburg
  - Skäne University Hospital, Lund
  - Södersjukhuset, Stockholm
  - Onkologikliniken, Uppsala